CLINICAL TRIAL: NCT05217914
Title: Copanlisib in Indolent Non-Hodgkin Lymphoma Patients: A Real-world Taiwan Observation Multicenter Study
Brief Title: A Study to Learn More About Copanlisib Treatment Patterns in People With Indolent Non-Hodgkin Lymphoma, a Type of Cancer That Grows and Spread Slowly and Develops in the Lymphatic System (a Part of Immune System) in Taiwan Under Real-word Conditions
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21960
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Relapsed or Refractory Indolent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence | interventions — copanlisib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- r/r iNHL Patients: Copanlisib treatment: The data in patients who received at least one dose of copanlisib before 01-May-2022 will be included for interim analysis. All study data collection will end in Q2 2024, or when the data collection of maximal 50 enrolled patients is completed, whenever comes first.
  Subgroup analysis: r/r iNHL Patients: Copanlisib 2nd line treatment Subgroup analysis: r/r iNHL Patients: Copanlisib 3rd line treatment
  Interventions: Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (BAY80-6946) — Copanlisib for treatment of relapse/refractory (r/r) indolent non-Hodgkin lymphoma (iNHL)

SUMMARY:
This is an observational study, in which data from Taiwanese people with indolent non-Hodgkin lymphoma who will be receiving copanlisib is studied.

Indolent non-Hodgkin lymphoma (iNHL) is a type of cancer that grows and spread slowly and begins in the lymphatic system, which is a part of body's immune system, and affects a type of white blood cells called lymphocytes of. In iNHL, white blood cells grow abnormally and can form growths (tumors) throughout the body. iNHL tends to come back after treatment (relapse) and may stop to respond to medical treatment (become refractory). While the disease is typically slow growing, it can become more aggressive over time. iNHL consists of multiple subtypes and it is already known to the researchers that Taiwanese people often have a different subtype of iNHL and poorer survival than people in most Western countries. Moreover, there is little information about how well the drug copanlisib works in Asian people with iNHL.

The study drug copanlisib works by blocking PI3K proteins and preventing cancer cells from growing and surviving. Copanlisib is already available in US and in Taiwan and is approved for doctors to prescribe to patients.

The National Authority for Health in Taiwan granted an accelerated approval of copanlisib due to the new mechanism of action of this drug and based on the results of a previous study, in which participants with iNHL received treatment with copanlisib. This previous study, however, included only a small number of Asian people and no Taiwanese people at all.

The main purpose of this study is to learn more about treatment patterns of copanlisib from Taiwanese people who have decided with their doctor to start copanlisib for iNHL.

To do this, researchers will collect the following data:

* administered doses of copanlisib
* dates of treatment administration
* how long copanlisib treatment was given
* the number of treatment periods also called cycles (one cycle is defined as 3 intravenous treatments in 3 of 4 weeks)
* dates and reasons of copanlisib treatment interruption
* dates and reasons of copanlisib treatment discontinuations. In addition, researchers will also look at how well copanlisib works in these people.

There are no required visits to the study site. The participants will receive their treatments as agreed with their doctors. The data will be gathered from the medical charts of the participants with iNHL who will receive copanlisib or received at least one dose of copanlisib after 01-Nov-2019. The data collection will cover the time between the date with the first diagnosis of iNHL and 01-May-2024 or earlier if the data collection of maximal 50 participants is completed before 01-May-2024.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of r/r iNHL
* Patients ages ≥ 18 years old when first dosed with copanlisib for iNHL.
* Patients who will receive copanlisib or received at least one dose of copanlisib after 01-Nov-2019
* Patients or his/her legal guardian or representative agree to provide the written informed consent or a waiver of informed consent granted by local IRB

Exclusion Criteria:

* Patients who had participated in the global clinical study for copanlisib before local market approval
* Patients who participate in an interventional trial during the data collection period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible r/r iNHL patients who will receive copanlisib or received at least one dose of copanlisib after 01-Nov-2019 and agreed to provide the written informed consent or a waiver of informed consent granted by local IRB.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Dose regimes | Approximately up to 27 month
  The treatment regimens of copanlisib including the reasons of copanlisib interruption within a cycle and discontinuation, if available, will be summarized by listing and presented as count and percentage if applicable.
Treatment duration | Approximately up to 27 month
  The treatment regimens of copanlisib including the reasons of copanlisib interruption within a cycle and discontinuation, if available, will be summarized by listing and presented as count and percentage if applicable.
Number of treatment cycles | Approximately up to 27 month
  The treatment regimens of copanlisib including the reasons of copanlisib interruption within a cycle and discontinuation, if available, will be summarized by listing and presented as count and percentage if applicable.
  Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle.
Reasons of discontinuations | Approximately up to 27 month
  The treatment regimens of copanlisib including the reasons of copanlisib interruption within a cycle and discontinuation, if available, will be summarized by listing and presented as count and percentage if applicable.

SECONDARY OUTCOMES:
Ann Arbor stage of the first diagnosis of iNHL | Approximately up to 27 month
Previous treatment regimens | Approximately up to 27 month
  Previous treatment regimens from the first diagnosis of iNHL until the initiation of copanlisib, including the duration from the first diagnosis of iNHL to the first dose of copanlisib, the POD (i.e., POD > 24 or POD ≤ 24) after the first line anticancer therapy for iNHL, and the duration from the most recent PD to the first dose of copanlisib.
Type of treatment response | From baseline to the end of each copanlisib treatment cycle (Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle)
  Type of treatment response [complete response (CR)/ complete response undefined (CRu)/partial response (PR)] based on the physicians' assessment according to local standard.
Duration of response (DoR) | From baseline to the end of each copanlisib treatment cycle (Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle)
Time to response | From baseline to the end of each copanlisib treatment cycle (Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle)
Progression status after the first dose of copanlisib | From baseline to the end of each copanlisib treatment cycle (Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle)
Time to progression | From baseline to the end of each copanlisib treatment cycle (Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle)
Largest change in target lesion size as judged by physicians | From baseline to the end of each copanlisib treatment cycle (Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle)
Number of patients with treatment-emergent AEs | Approximately up to 27 month
Change in laboratory data, including hemoglobin A1c (HbA1c) values | From baseline to the end of each copanlisib treatment cycle (Three intravenous infusions of copanlisib dosing in a 28-day intermittent treatment schedule (i.e., 3 weeks on and 1 week off) will be regarded as a treatment cycle)
Subsequent therapeutic options for treating iNHL post discontinuation of copanlisib | Approximately up to 27 month

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com